CLINICAL TRIAL: NCT06654037
Title: A Phase 1 Study of 5-Fluorouracil in Combination With Abemaciclib in Metastatic, Refractory CRC
Brief Title: Testing the Addition of an Anti-Cancer Drug, Abemaciclib, to the Usual Chemotherapy Treatment (5-Fluorouracil) for Metastatic, Refractory Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-08691; NCI-2024-08691 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10670 (Other: UPMC Hillman Cancer Center LAO); 10670 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Microsatellite Stable Colorectal Carcinoma; Refractory Microsatellite Stable Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — abemaciclib; Biopsy; Specimen Handling; Fluorouracil; dehydroftorafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (abemaciclib, 5-FU) (Experimental): Patients receive abemaciclib PO BID on days 1-28 and 5-FU IV over 46 hours on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and radiologic imaging throughout the study and may additionally undergo a tissue biopsy before treatment and on cycle 1 day 16.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Fluorouracil; Procedure: Radiologic Imaging Procedure

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Procedure: Radiologic Imaging Procedure — Undergo radiologic imaging

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of abemaciclib in combination with 5-fluorouracil and how well it works in treating patients with colorectal cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and that has not responded to treatment (refractory). Abemaciclib, a type of cyclin-dependent kinase inhibitor, blocks certain proteins, which may help keep tumor cells from growing. 5-fluorouracil, a type of antimetabolite, stops cells from making deoxyribonucleic acid (DNA) and may kill tumor cells. Giving abemaciclib in combination with 5-fluorouracil may be safe, tolerable, and/or effective in treating patients with metastatic and refractory colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of abemaciclib in combination with 5-fluorouracil (5-FU) in patients with colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To estimate the anti-tumor activity of abemaciclib in combination with 5-FU. II. To determine the pharmacodynamics (PD) of abemaciclib in combination with 5-FU (death receptor 5 [DR5] dynamics and apoptosis).

III. To identify molecular subpopulations particularly sensitized to abemaciclib and 5-FU.

IV. To determine the pharmacokinetics (PK) of abemaciclib and 5-FU.

EXPLORATORY OBJECTIVES:

I. To explore exposure-response relationships for abemaciclib and 5-FU. II. To evaluate circulating tumor DNA (ctDNA) as a predictor for treatment response to therapy.

OUTLINE: This is a dose-escalation study of abemaciclib in combination with 5-FU followed by a dose-expansion study.

Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-28 and 5-FU intravenously (IV) over 46 hours on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and radiologic imaging throughout the study and may additionally undergo a tissue biopsy before treatment and on cycle 1 day 16.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed microsatellite stability (MSS) metastatic colorectal cancer where patients have progressed on standard therapies which would have included 5-FU or capecitabine, oxaliplatin, and irinotecan. Patients must have had progression of disease (PD) or intolerance to bevacizumab and anti-EGFR antibodies (cetuximab or panitumumab) in patients who have left-sided and RAS-wildtype colorectal cancer (CRC)
* Patients must have measurable disease
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of abemaciclib in combination with 5-FU in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN for patients who do not have liver metastases, and ≤ 5 x institutional ULN for patients with liver metastases
* Glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patients must have available archival tumor tissue at the time of patient enrollment for molecular profiling studies. A biopsy may be done if archival tissue is not available
* Palliative radiation for symptom management to a metastatic site will be permitted during the course of the study. Please discuss specific cases with the national principal investigator (PI)
* Patients must have completed previous systemic therapy for at least five half-lives or 2 weeks, whichever is shorter, prior to study dosing
* Patients who have not had major surgery within 14 days prior to randomization
* Patients who do not have serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance < 30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea)
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization
* Patients who are able to swallow oral medications
* Patients who do not have a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Patients who do not have an active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment) or fungal infection
* The effects of abemaciclib on the developing human fetus are unknown. For this reason and because cyclin-dependent kinases (CDK) inhibiting agents as well as other therapeutic agents used in this trial are known to be teratogenic, men and women treated or enrolled on this protocol must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to the study, for the duration of study participation, and 3 months after completion of abemaciclib and fluorouracil. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia or grade 2 peripheral neuropathy. Patients who are experiencing immune related adverse events (AEs) which are adequately treated with hormone replacement therapy, including diabetes on insulin regimen, hypothyroidism on levothyroxine, and adrenal insufficiency on steroid replacement will also be eligible
* Patients who are receiving any other investigational agents. There is to be a washout period of two weeks or five half-lives, whichever is shorter, for all investigational agents prior to treatment initiation on this study. Individual cases can be discussed with the national PI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib or other agents (5-FU) used in study such as a previous intolerance to 5-FU or capecitabine, including patients with known or suspected dihydropyrimidine dehydrogenase deficiency
* Patients who have received previous treatment with a CDK4/6 inhibitor
* Patients with a gastrointestinal pathology or history that adversely impacts the ability to take or absorb oral medication
* Patients with peritoneal metastases complicated by ascites which are refractory to diuretic therapy and requires therapeutic paracenteses more than once every 2 weeks
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A enzymes before enrollment or while on protocol therapy are ineligible. Patients receiving moderate CYP3A inhibitors or inducers will be monitored. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because abemaciclib is a CDK-inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with abemaciclib, breastfeeding should be discontinued if the mother is treated with abemaciclib. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within first cycle (cycle length = 28 days)
  Will be tabulated using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 for each dose level.
Maximum tolerated dose (MTD) | Up to completion of dose-escalation phase
  MTD will be the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate.
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Will be evaluated using CTCAE v 5.0 and will be tabulated for each dose level.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months post-treatment
  ORR will be defined as the addition of complete response and partial response. Response will be assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. The probability of ORR will be estimated with exact 95% binomial confidence intervals.
Clinical benefit rate | Up to 6 months post-treatment
  Will be assessed using RECIST v 1.1.
Progression free survival (PFS) | From the start of treatment to time of progression or death up to
  PFS will be assessed using the Kaplan-Meier method, along with 95% confidence interval.
Ribonucleic acid sequencing of death receptor 5 | At pre-treatment on cycle 1 day 16
  Pre-post comparisons will be made within patients being biopsied, using a non-parametric paired test, at a significance level (alpha) of 0.05.
Apoptosis by Pharmacodynamics Assay Development & Implementation Section lab | At pre-treatment cycle 1 day 16
  Pre-post comparisons will be made within patients being biopsied, using a non-parametric paired test, at a significance level (alpha) of 0.05.
Whole exome sequencing of archival tissue | Up to cycle 1 day 1 pre-dose
  Will look for mutations in genes relevant to deoxyribonucleic acid (DNA) damage repair, signaling and (fluoropyrimidine) metabolism and in a descriptive manner evaluate any relations with peculiar response and/or toxicity.
Pharmacokinetics (PK) of abemaciclib and possibly active metabolites M2, M20, and M18 in plasma and tumor tissue | At pre-dose on cycle 1 days 1, 2, 8, and 15 and at cycle 2 days 1 and 15
  Abemaciclib PK will be evaluated and compared descriptively with historical data.
PK of 5-fluorouracil (5-FU) | At cycle1 day 1 pre-dose and cycle 1 day 2 (22-26 hours post start of 5-FU infusion)
  Will be evaluated by area under the concentration-time curve (AUC) and be compared descriptively with historical data.

OTHER OUTCOMES:
Abemaciclib AUC and trough levels 5-FU AUC | At cycle1 day 1 pre-dose and cycle 1 day 2 (22-26 hours post start of 5-FU infusion)
  Will be exploratorily correlated with toxicity and response with non-parametric tests at a significance level of 0.05 (PK endpoints in patients with versus without presence of toxicity or response endpoints). Abemaciclib tissue exposure and tissue to plasma ratios will be descriptively reported.
Change in variant allele frequencies (VAF) of tumor mutations in circulating tumor DNA | At baseline and at start of cycle 3 (cycle length = 28 days)
  The detectable VAFs will be assessed and trended during the course of treatment. VAF change will be assessed categorically for each patient (increased or decreased at start of cycle 3 as compared to baseline). The association of VAF change with objective response will be tested using the Fisher's test, where p < 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Janie Y Zhang, Principal Investigator — UPMC Hillman Cancer Center LAO
Locations (8):
- United States (8):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm